CLINICAL TRIAL: NCT05106699
Title: Carbon Ion Boost Followed by Pelvic Proton Radiotherapy for Prostate Cancer With Pelvic Lymph Nodes Metastases: Prospective Phase II Study
Brief Title: Carbon Ion Followed by Proton Radiotherapy for Prostate Cancer With Pelvic Lymph Nodes Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Ping Li, Associate chief physician, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-PCa2021-01
Record Dates: First submitted 2021-10-24; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
Keywords: Carbon ion; Proton; prostate cancer; pelvic lymph nodes metastases
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Protons

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carbon ion followed by Proton radiotherapy (Experimental): All patients received whole pelvis and prostate region radiotherapy. The dose to metastatic LN was escalated using simultaneous integrated boost (SIB) technique.
  Interventions: Radiation: proton plus carbon ion radiation

INTERVENTIONS:
Radiation: proton plus carbon ion radiation — All patients received whole pelvis and prostate region proton irradiation of 46 GyE in 23 fractionsfollowed by localized carbon ion irradiation of 32GyE in 8 fractions to the prostate region. The dose to metastatic LN was escalated using simultaneous integrated boost (SIB) technique. The dose was 60-62.1GyE in 23 fractions as much as dose constraints. All patients will be recommened receive 2-3 years endocrine therapy.

SUMMARY:
The present of clinically pelvic lymph node positive (cN1) represent one of the most important prognostic factors for recurrence and cancer-specific mortality of prostate cancer patients. Approximately 12% of prostate cancer patients present with cN1 disease at the time of diagnosis. Furthermore, with the advent of more sensitive advance diagnostic imaging techniques, such as PSMA PET/CT, the likelihood that pelvic nodes will be found earlier and more frequently.

Unfortunately, The optimal treatment for patients with cN1 still remains unclear. Androgen deprivation therapy (ADT) is the cornerstone of prostate cancer with pelvic lymph node metastasis. Some retrospective and database studies have shown that addition of local radiotherapy (RT) to ADT improve the treatment outcome. The 2022 NCCN guideline recommend RT combined with 2 to 3 years ADT in patients with initially diagnosed cN1 prostate cancer who have a life expectancy greater than 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven initial diagnosis of adenocarcinoma of the prostate;
* Clinical stage T1-4 N0 M0;
* Prostatic assessment by multiparametric (mp) MRI;
* Pelvic lymph node was assessed by PSMA PET/CT and mpMRI;
* No distant metastasis was proven by PSMA PET/CT;
* Patients may received neoadjuvant hormonal therapy;
* 45≤ Age ≤85;
* Adequate performance status (ECOG 0-1);
* No previous pelvic radiation therapy (RT);
* No previous prostatectomy;
* No previous invasive cancer (within 5 years before the prostate cancer diagnosis);
* Ability to understand character and individual consequences of the clinical trial;
* Written informed consent;

Exclusion Criteria:

* No pathologically confirmed adenocarcinoma of the prostate;
* Distant metastasis (M1);
* Previous pelvic radiotherapy;
* Previous prostatectomy;

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical relapse free survival | From the start of systemic therapy, a median of 3 years
  The prostate specific antigen less than nadir plus 2ng/ml (Phoenix definition)

SECONDARY OUTCOMES:
Progression free survival | From the start of systemic therapy, a median of 3 years
  The time from start of systemic therapy to tumor progression or death
Overall survival | From the start of systemic therapy, a median of 3 years
  The time from diagnosis to death from any cause
Metastasis free survival | From the start of systemic therapy, a median of 3 years
  The time from start of systemic therapy to tumor metastatsis.
Acute toxicities | Within 3 months of the start of particle therapy
  Treatment related acute toxicity assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Late toxicities | 3 months after the completion of particle therapy
  Treatment related late toxicity assessed by Radiation Therapy Oncology Group (RTOG) scale

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhang, M.D., Study Director — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, China